CLINICAL TRIAL: NCT00509548
Title: An Open-Label Randomized Pilot Study of Safety and Preliminary Efficacy of TG100801 in Patients With Choroidal Neovascularization Due to Age-Related Macular Degeneration
Brief Title: Open-Label, Pilot Study of TG100801 in Patients With Choroidal Neovascularization Due to AMD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: TargeGen (Industry)
Responsible Party: Jolene Shorr/Senior Director, Clinical Development, TargeGen, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH-TG100801-002
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Macular Degeneration; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — 4-chloro-3-(5-methyl-3-((4-(2-pyrrolidin-1-ylethoxy)phenyl)amino)-1,2,4-benzotriazin-7-yl)phenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Dose 1
  Interventions: Drug: TG100801
- 2 (Experimental): Dose 2
  Interventions: Drug: TG100801

INTERVENTIONS:
Drug: TG100801 — Eye drop, twice a day, 30 days.

SUMMARY:
Wet age-related macular degeneration (AMD) is caused by the formation and growth of abnormal blood vessels (angiogenesis) in the retina. The new blood vessels have fragile walls and can leak fluid into the retina. The build-up of fluid (edema) under the macula can distort vision or cause vision loss. TG100801 is a topical (eye drop) therapy that has been shown to inhibit ocular angiogenesis, vascular leak, and inflammation in laboratory studies. The primary purpose of this pilot study is to evaluate the ability of topical administration of TG100801 to reduce the amount of fluid in the retina in patients with AMD following 30 days of treatment. An additional objective is to evaluate the safety of TG100801 in patients with AMD.

DETAILED DESCRIPTION:
Choroidal neovascularization (CNV) due to AMD is the leading cause of irreversible, severe vision loss in people 55 years and older in the developed world. TG100801 is a potent inhibitor of vascular growth endothelial factor (VEGF) and other kinases that contribute to CNV and macular edema. Animal models have demonstrated the ability of TG100801 to inhibit angiogenesis, vascular leak, and inflammation. TG100801 is being developed as a topical (eye drop) therapy for treatment of CNV due to AMD.

The primary objective of this multicenter, open-label, randomized, pilot study is to evaluate the effects of 30 days of dosing with two dose levels of TG100801 on central retinal/lesion thickness, as measured by optical coherence tomography (OCT). The safety of TG100801 in patients with AMD also will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal CNV secondary to AMD in study eye
* CNV lesion size less than or equal to 12 MPS disk areas
* CNV > 50% of lesion area
* Presence of intraretinal fluid causing an increase in central subfield thickness of at least 250 microns, confirmed by OCT in study eye
* Any lesion composition
* Best corrected visual acuity of 20/40 to 20/320 (73 to 24 ETDRS letters) at 4 meters in study eye
* Best corrected visual acuity of 20/800 or better (at least 4 ETDRS letters) at 4 meters in fellow eye
* Ability to administer and tolerate eye drops
* Able to give written informed consent

Exclusion Criteria:

* History of any treatment for subfoveal CNV in study eye
* Known or anticipated need for use of topical medication in study eye during 30-day dosing period
* Current or anticipated need for any available ocular anti-VEGF therapy in fellow eye for 30 days prior to and 30 days following baseline
* RPE rip or tear in study eye
* Blood > 1 disk area, atrophy, or fibrosis (disciform scar) under foveal center of study eye
* Scarring/fibrosis of at least 25% of total CNV lesion in study eye
* Hemorrhage or PED > 50% of total CNV lesion in study eye
* Glaucoma with visual field loss or IOP at least 25 mmHg in study eye or consistently at least 25 mmHg in fellow eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in central retinal/lesion thickness as measured by OCT at Week 4. | 4 weeks

SECONDARY OUTCOMES:
Mean/median change in visual acuity from baseline. Proportion of subjects with loss of > 15 ETDRS letters. Proportion of subjects with loss of > 30 ETDRS letters. Proportion of subjects gaining at least 15 letters. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kaiser, M.D., Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (8):
  - Retina Centers, PC, Tucson, Arizona
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Vitreous-Retina-Macula Consultants of New York, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Vitreoretinal Consultants, Houston, Texas

REFERENCES:
- See also: American Macular Degeneration Foundation — http://www.macular.org